CLINICAL TRIAL: NCT04984265
Title: Noninvasive Cardiac Radiation for Ablation of Ventricular Tachycardia in Chagas Disease Patients
Brief Title: SBRT in Chagas Disease Ventricular Tachycardia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Mauricio Ibrahim Scanavacca, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4920/19/139
Record Dates: First submitted 2021-07-21; First posted 2021-07-30 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Ventricular Tachycardia; Chagas Disease; Cardiac Arrhythmia
Keywords: Cardiac Radioablation; Chagas Disease; Refractory Ventricular Tachycardia; Stereotactic Body Radiation Therapy; SBRT
MeSH Terms: conditions — Tachycardia, Ventricular; Chagas Disease; Arrhythmias, Cardiac | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Body rRadiotherapy (SBRT) (Experimental): SBRT targeting the area of the circuit of Ventricular Tachycardia
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — SBRT targeting the area of the circuit of Ventricular Tachycardia
  Other Names: SBRT

SUMMARY:
This is an observational study of 10 Chagas Disease patients with Ventricular Tachycardia that have failed prior catheter ablation or have this procedure contraindicated due to clinical status. Those patients will underwent to Stereotactic Body Radiation Therapy (SBRT) targeting the area of the heart of the VT circuits. Radioablation target will be defined based on prior ablation electroanatomical mapping, VT morphology, pre-acquired imaging (CT angiogram, Cardiac Magnetic Resonance), current imaging reconstructed and integrated to electroanatomical mapping and a EP study to define current VT morphologies. Gross targeted volume (GTV), internal targeted volume (ITV) and planning targeted volume (PTV) will be defined and calculated and a single 25Gy dose will be delivered to the PTV. Patients will be followed initially for one year and efficacy endpoint will be rate of VT recurrence, time to recurrence and VT burden. Safety endpoint will be the occurrence of any adverse effect related to SBRT.

DETAILED DESCRIPTION:
Enrollment A patient that fulfill all inclusion criteria (especially diagnosis of Chagas heart disease including positive serology, recurrent sustained ventricular tachycardia requiring therapy and failed or is ineligible for catheter ablation and had no exclusion criteria will be identified as a candidate for participation in this study while receiving care at Instituto do Coração, São Paulo, Brazil. The clinical team will contact the patient in-person and propose study participation and Consent Form will be applied.

A total of 10 patients will be enrolled in the current study. At the time of enrollment, baseline information pertaining to symptoms and details regarding clinical presentation, imaging, and heart catheterization procedures will be obtained from examination of their medical record and recorded in a Redcap database.

Pre-radiation Imaging and Definition of Treatment Area:

All patients will perform a cardiac MRI with 3D LGE sequence to be imported in the ADAS 3D software. After MRI acquisition, images will be imported in the software, segmented and the channels will be identified using an specific tool in the software. After channels and scar identified the quality of reconstruction and channel identification will be manually validated by one of the investigators. If the image is considered adequate, the scar, the chambers and the channels will be exported in VTK format. If the reconstruction is defined as a poor quality by the investigators, last VT ablation procedure and or ECGs of the VT and cardiac, mapping data from prior ablation, prior MRI or cardiac CT analyzing wall thickness will be used to design treatment area . Additionally, areas of scar or infarction identified by previous electroanatomic mapping (voltage maps), imaging (CT, echocardiography, and/or nuclear imaging) that are likely the source of VT based on mapping or ECG analysis will be targeted. The area of interest will be determined by both the treating cardiologist and radiation oncologist.

Radiation treatment:

Simulation:

All patients will undergo a 4D CT scan for treatment planning. The patient will be immobilized using a custom BodyFIX device. CT with contrast is preferred to facilitate anatomical definition when the patient is a candidate for contrast.

Definition of the target volume:

As described above, the gross target volume (GTV) will be defined using the pre-radiation imaging. Using the 4D CT data, an internal target volume (ITV) will then be created to account for organ motion. Finally, to account for any patient setup variability, a planning target volume (PTV) will be created by adding a 5 mm margin to the ITV. The prescribed dose will be 25 Gy to the PTV.

The following are recommendations for radiation planning parameters with regards to target coverage and normal tissue constraints. Final determination regarding radiation treatment plan approval is left at the treating provider's discretion.

Treatment planning guidelines:

* 95% of the PTV should be covered with 100% of the prescribed dose
* 100% of the ITV should be covered with 100% of the prescribed dose Dmax of 120% the prescribed dose SBRT will take place at the radiation oncology department. Treatment will be completed within approximately 90 minutes during one visit.

Post ablation management Any ICD or pacemaker will be interrogated before and immediately after ablation and settings and function documented. Continued antiarrhythmic drug therapy will be left to the discretion of the treating physicians. The following approaches are recommended: If the patient is receiving amiodarone, it is recommended that the dose be reduced to 200 mg daily and then consider stopping it after 3 months if no VT has occurred in the previous month. It is recommended that antiarrhythmic drugs combined with amiodarone be stopped at 6 weeks after radioablation if VT has not recurred in the preceding two weeks. For other antiarrhythmic medications in the absence of amiodarone, continuing administration for the first 3 months is recommended if tolerated.

Anticoagulation with warfarin or a direct acting anticoagulant will be maintained for one month.

Follow-up Follow up will be at 4-6 weeks, 10-14weeks, 5-7 months, 11-13 months and thereafter every 1 year. At the above intervals, all patients will return for follow-up in the Department of Cardiology and Department of Radiation Oncology. At each visit screening for effectiveness and adverse effects attributable to treatment will be performed. Arrhythmia burden will be determined from ICD interrogation. Ventricular function will be assessed from echocardiography at 3 months. Side effects will be graded according to CTCAE v4.0 criteria.

Patients who die during the follow-up period will be considered for autopsy to evaluate the effect of treatment at the histologic and cellular level. This will be subject to approval by the patient or his/her family.

Risks The principal elements of risk in the study are possible complications of ablative doses of radiation targeting the ventricle. Target regions and radiation doses will be designed to limit dose to surrounding normal tissues using established constraints to minimize potential toxicity. Treatment experience for an electrically ablative dose of radiation to the myocardium is based on case reports and series noted above. Potential side effects include, but are not limited to, skin changes/fibrosis, rib weakening or fracture, lung injury (pneumonitis or fibrosis), heart injury (decreased EF, pericarditis, or conduction abnormalities), vascular injury (to coronaries or other major vessels), nerve or spinal injury, esophageal injury (stricture or esophagitis), fatigue, birth defects, and secondary malignancy.

Given the severe detriment to quality of life and survival in patients with recurrent VT and the evidence of VT burden reduction in patients treated with stereotactic ablation, we believe the benefits of further characterizing this technique justify the risks.

Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others Any unanticipated adverse events will be reported by the Principal Investigator according to applicable IRB policy. The PI is fully engaged in the actual performance of the study and this ensures that adverse events would be readily known and reported by the PI.

Study Withdrawal/Discontinuation If an individual decides to withdraw their consent by informing study staff in writing or verbally, we will withdraw the participant. Contact information for the PI and study staff will be made available to the participant upon enrollment in the consent document.

Data Management Data will be stored in REDCap using the participant's study ID. Their REDCap data record may contain some identifying information. Subjects will be tracked using their study ID. The identifiable data, excluding date of procedures, will reside as a separate form under the data entry sections labeled "Registration/PHI" within our REDCap database which will allow us to exclude access to the identifiable information, excluding date of procedures, if necessary. Minimal paper records will be kept, and they will be kept locked in a cabinet.

Study protocol will adhere to privacy regulations at Instituto do Coração. No information will be released, nor will participation in the research be acknowledged, to any party except where compulsory according to law or Instituto do Coração policy. There may be unknown or unanticipated adverse effects from participation in this registry for which the PI and study team will remain observant.

12. Follow-up and Record Retention Patient will be enrolled until the number is complete. Data will be retained indefinitely. Electronic data may be destroyed earlier at the request of the participant. Electronic records will be deleted from the REDCap database, paper copies will be deposited into locked containers designated for shredding of confidential patient information.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Chagas heart disease including positive serology
2. Recurrent sustained ventricular tachycardia requiring therapy due to symptoms, ICD shocks, or requiring hospitalization.
3. Age>18 years.
4. Able to give written, informed consent. If the patient requires continuous sedation/anesthesia for arrhythmia control consent can be provided by the next of kin.
5. Medically fit to undergo radiation planning and treatment sessions.
6. Failed antiarrhythmic medications due to VT recurrence, drug intolerance, or contraindication.
7. Failed prior catheter ablation due to arrhythmia recurrence or ineligible for endocardial or epicardial catheter ablation (LV thrombus, epicardial adhesion, megacolon, prior open chest surgery)

Exclusion Criteria:

1. Cardiogenic shock not due to VT with no possibility of heart transplant or ventricular assist device.
2. Inability for patient to be adequately immobilized for radiation planning and treatment.
3. Repeat catheter ablation is felt to be a reasonable option.
4. Previous radiation to the chest.
5. Pregnancy or refusal to use contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety of SBRT for the treatment of Ventricular Tachycardia | 12 months
  Incidence of cardiac and extra-cardiac adverse effects related to SBRT
Efficacy of SBRT for the treatment of Ventricular Tachycardia | 12 months
  Rate of VT recurrence after a blanking period of 6 weeks following SBRT

SECONDARY OUTCOMES:
Time to VT Recurrence | 12 months
  Time to VT recurrence after a blanking period of 6 weeks following SBRT
VT Burden | 12 months
  Number of ICD therapies following SBRT compared to 12 months before
Mortality | 12 months
  Rate of mortality following SBRT
Cardiac Mortality | 12 months
  Rate of mortality due to cardiac causes following SBRT

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio I Scanavacca, MD, PhD, Study Director — University of São Paulo General Hospital
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil